CLINICAL TRIAL: NCT03112057
Title: Visualize Nociceptor Changes in Neuropathic Human
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201610037DINC
Record Dates: First submitted 2017-03-28; First posted 2017-04-13 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-03

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy subjects (Experimental): Healthy subjects of different ages (20 persons), Interventions: harmonic generation microscopy
  Interventions: Diagnostic Test: harmonic generation (HGM) microscopic methods.
- peripheral neuropathy (Experimental): the participant have symptoms and diagnosed with peripheral neuropathy (90 persons), Interventions:harmonic generation microscopy
  Interventions: Diagnostic Test: harmonic generation (HGM) microscopic methods.
- diabetic neuropathy (Experimental): the participant have symptoms and diagnosed with diabetic neuropathy (20 persons), Interventions:harmonic generation microscopy
  Interventions: Diagnostic Test: harmonic generation (HGM) microscopic methods.
- chemotherapy induced neuropathy (Experimental): before chemotherapy, during chemotherapy, after peripheral nerve lesions were cured (30 persons). Interventions:harmonic generation microscopy
  Interventions: Diagnostic Test: harmonic generation (HGM) microscopic methods.
- Polydactyly (Experimental): Abandoned extra digit specimen of polydactyly(10 persons): the normal skin and nerve endings in extra digit: Interventions: harmonic generation microscopy
  Interventions: Diagnostic Test: harmonic generation (HGM) microscopic methods.

INTERVENTIONS:
Diagnostic Test: harmonic generation (HGM) microscopic methods. — a frequency-dependent optical microscopy system with a near-infrared light source with a wavelength of 1230 nm was used to detect the diseased site and normal skin.Use erbium-Jacob (Er-YAG) laser exfoliation. the participants need to lie down, wear goggles. The lens sucker device to help fix the skin examination site. Based on the experience of the past 118 subjects, the participants did not discomfort. The total time of the laser irradiation on the same skin is no more than 30 minutes, the maximum laser power is no more than 0.15 watts, irradiation in the skin of the total energy of the laser does not exceed 270 joules. After the experiment, the investigators immediately check the skin for the participants

SUMMARY:
The purpose of this experiment is to establish a solid medical foundation for the successful development of non-invasive harmonic generation (HGM) microscopic slicing methods. The purpose of this new technology platform is to directly observe the nerve endings of nociceptors To enhance understanding of how neuropathies occur, persistence, and ease. This technique will assist in the diagnosis and prognosis of patients with neuralgia.

DETAILED DESCRIPTION:
This study will be the skin tissue for the virtual slice object, the study intends to the following research:

The number of people enrolled in the Court is 170.

Between 20 and 90 years old, meet the following conditions, suitable for participation in this test:

1. Healthy subjects of different ages (20 persons): to study the optical imaging of the skin and nerve endings: the control of healthy subjects and peripheral neuropathy patients skin observed by the optical images of the shoots.
2. Abandoned extra digit specimen of polydactyly(10 persons): to study the optical imaging of the normal skin and nerve endings in extra digit : collect abandoned digit specimen after surgical removal in polydactyly.
3. has been diagnosed with peripheral neuropathy (90 persons):to study the diagnosis of peripheral neuropathy of the skin nerve endings of the optical image observation and quantitative sensory nerve examination
4. clinically must be diagnosed by the skin slices of diabetic neuropathy patients have been removed after the completion of clinical diagnosis of the specimen,And then the skin slices of the nerve endings of the optical image observation (20 persons):study the technical observation of diabetic patients with skin sections of the nerve endings of the optical image observation: the clinical must be skin slices for the diagnosis of diabetic neuropathy, patients has been taken out after the completion of clinical diagnosis, and then the skin slices of the nerve endings of the light learning image observation.
5. because of chemotherapy during chemotherapy, is expected to have peripheral neuropathy: before the occurrence of peripheral neuropathy , Peripheral nerve lesions were cured after subcutaneous nerve optical observation (30 persons):for different periods of peripheral neuropathy subcutaneous nerve optical observation: in the peripheral neuropathy occurred before the occurrence of peripheral neuropathic symptoms, peripheral neuropathy after cure for subcutaneous nerve optical observation.

This test can not be attended if:

Those who suffer from systemic infection or have been infected with the site by the physician assessment is not suitable for examination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects of different ages
* abandoned extra digit specimen in polydactyly
* diagnosed with peripheral neuropathy
* diabetic neuropathy patients have been removed after the completion of clinical diagnosis of the specimen, And then the skin slices of the nerve endings of the optical image observation
* because of chemotherapy during chemotherapy, is expected to have peripheral neuropathy: before the occurrence of peripheral neuropathy , after cured peripheral nerve lesions

Exclusion Criteria:

* systemic infection or have been infected with the site by the physician assessment is not suitable for examination.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
nerve ending number measurement | through study completion, an average of 1 year
  Use of harmonic generation (HGM) microscopic virtual biopsy methods to obtain 3D live images.

SECONDARY OUTCOMES:
nerve ending structure measurement | through study completion, an average of 1 year
  Quantify the molecules on the image, the biological characteristics of tissue nerve cells have a comprehensive understanding, and will try to establish the human subcutaneous nerve optical observation method

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan